CLINICAL TRIAL: NCT02159664
Title: Influence of Didgeridoo Practice on Upper Airways Obstruction Levels in Moderate Obstructive Sleep Apnea Patients
Brief Title: Influence of Didgeridoo Practice on UA Obstruction Levels in Moderate OSA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty to recrut patients
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Principal Investigator, Marie Bruyneel, Influence of didgeridoo pratice on upper airways obstruction levels in moderate obstructive sleep apnea patients, Centre Hospitalier Universitaire Saint Pierre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK/14-03-25/4354
Record Dates: First submitted 2014-06-06; First posted 2014-06-10 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Sleep Apnea
Keywords: didgeridoo; sleep apnea; drug induced sleep endoscopy
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- didgeridoo practice (Experimental)
  Interventions: Other: didgeridoo practice

INTERVENTIONS:
Other: didgeridoo practice — instrument lessons, 1X/w and daily practice, 20 min /d

SUMMARY:
Didgeridoo practice has been shown to improve OSA severity. The aim of our study is to assess the changes in upper airways obstruction levels before and after Didgeridoo practice in moderate OSA patients.

DETAILED DESCRIPTION:
Didgeridoo practice has been shown to improve Obstructive Sleep Apnea (OSA) severity. The aim of our study is to assess the changes in upper airways obstruction levels, evaluated by sleep endoscopy, before and after 3 months of Didgeridoo practice in moderate non obese OSA patients. Severity of OSA will also be documented by polysomnography.

ELIGIBILITY:
Inclusion Criteria:

* moderate OSA, non obese

Exclusion Criteria:

* not willing play didgeridoo age<18 significant lung, cardiac disease neuromuscular disease psychiatric disorders drugs with influence on respiratory drive

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-12; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
upper airways obstruction levels | 3 months
  assessed by drug-induced sleep endoscopy

SECONDARY OUTCOMES:
apnea-hypopnea index | 3 months
  assessed by polysomnography

OTHER OUTCOMES:
subjective sleep quality and sleepiness | 3 months
  assessed by questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Marie Bruyneel, MD, Principal Investigator — CHU St Pierre
Locations (1):
- CHU St Pierre, Brussels, Belgium